CLINICAL TRIAL: NCT04274764
Title: Sustainable Community Clinic Telemedicine-Based Glaucoma Screening
Brief Title: Screening and Intervention for Glaucoma and Eye Health Through Telemedicine
Acronym: SIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paula Anne Newman-Casey, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00169371; 5-U01-DP-006442-05-00 (Other Grant/Funding Number: Centers for Disease Control and Prevention); 5U01DP006442-05 (NIH)
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Glaucoma
Keywords: Telemedicine; Motivational interviewing; Health Coaching
MeSH Terms: conditions — Glaucoma | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Participants will be assigned at a 1:1 ratio to the study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized eHealth Education & Motivational Interviewing (Experimental): Personalized eHealth Glaucoma Education & Motivational Interviewing
  Interventions: Behavioral: Personalized eHealth Education & Motivational Interviewing
- Standard Education (No Intervention): Participant will receive standard glaucoma education.

INTERVENTIONS:
Behavioral: Personalized eHealth Education & Motivational Interviewing — This intervention uses a web-based application to generate personalized education materials for patients based on their eye health screening results and barriers to follow up care. A glaucoma counselor trained in brief, glaucoma-specific motivational interviewing (MI) uses the individualized content generated from this web-based application to form the basis of her conversation with the patient to coach the patient to engage in follow-up care.
  Arms: Personalized eHealth Education & Motivational Interviewing

SUMMARY:
This is a multiple site, randomized study that will assess the effects of personalized eHealth education and motivational-interviewing-based counseling on patient adherence to physician follow-up appointments.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effects of personalized eHealth education and motivational-interviewing-based counseling on adherence to glaucoma follow-up care compared to standard education delivered by a trained staff member. Participants will be randomized in a 1:1 ratio to either standard education and care navigation or eHealth education, counseling and care navigation. The outcome measure of the participant seeing an Ophthalmologist for follow up care within 3 months was increased to 6 months. This modification was made due to ophthalmology visit appointments not being available within the 3-month timeframe.

This study is embedded in a CDC-funded program to engage people from medically underserved areas in glaucoma screening. Participants who screened positive for glaucoma or suspected glaucoma were randomized in a 1:1 ratio to either the standard education and care navigation arm or the eHealth education, counseling, and care navigation arm.

ELIGIBILITY:
Inclusion Criteria:

- > or = to 18 years of age

Exclusion Criteria:

* Sudden vision changes
* Significant eye pain
* Pregnant women
* Prisoners
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Anne Newman-Casey, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Hamilton Community Health Clinic, Flint, Michigan
  - Hope Clinic, Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Newman-Casey PA, Killeen O, Miller S, MacKenzie C, Niziol LM, Resnicow K, Creswell JW, Cook P, Heisler M. A Glaucoma-Specific Brief Motivational Interviewing Training Program for Ophthalmology Para-professionals: Assessment of Feasibility and Initial Patient Impact. Health Commun. 2020 Feb;35(2):233-241. doi: 10.1080/10410236.2018.1557357. Epub 2018 Dec 20. PMID 31878800
- [Derived] Flaharty K, Niziol LM, Woodward MA, Elam A, Bicket A, Killeen OJ, Zhang J, Johnson L, Kershaw M, John DA, Wood SK, Musch DC, Newman-Casey PA. Association of Contrast Sensitivity With Eye Disease and Vision-Related Quality of Life. Am J Ophthalmol. 2024 May;261:176-186. doi: 10.1016/j.ajo.2024.01.021. Epub 2024 Jan 26. PMID 38281569
- [Derived] Newman-Casey PA, Aliancy J, Lu MC, Woodward MA, Hicks PM, Niziol LM, Musch DC, Bicket AK, John D, Killeen O, Wood SD, Johnson L, Kershaw M, Zhang J, Elam AR. Social Deprivation and the Risk of Screening Positive for Glaucoma in the MI-SIGHT Telemedicine-Based Glaucoma Detection Program. Ophthalmology. 2023 Oct;130(10):1053-1065. doi: 10.1016/j.ophtha.2023.05.021. Epub 2023 May 19. PMID 37211338
- See also: Hope Clinic — https://thehopeclinic.org/
- See also: Hamilton Clinic — https://www.hamiltonchn.org/main-clinic/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Personalized eHealth Education & Motivational Interviewing | Standard Education
Started | 309 | 313
Completed (Date of followup visit with an ophthalmologist was scheduled for a date prior to trial stop date) | 247 | 243
Not Completed | 62 | 70
Not completed — Date of scheduled followup visit was after trial stop date | 62 | 70

BASELINE CHARACTERISTICS:
Population: All participants are included whose date of followup visit with an ophthalmologist was scheduled for a date prior to trial stop date, and therefore whose outcomes could be assessed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized eHealth Education & Motivational Interviewing | Standard Education | Total
Number analyzed (Participants) | 247 | 243 | 490
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (14.2) | 58 (14.8) | 58.4 (14.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 95 | 88 | 183
  Female | 149 | 152 | 301
  Unknown/Refused/Prefer not to answer | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 200 | 194 | 394
  Unknown or Not Reported | 39 | 43 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 164 | 165 | 329
  White | 62 | 49 | 111
  More than one race | 7 | 10 | 17
  Unknown or Not Reported | 10 | 9 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 247 | 243 | 490

OUTCOME MEASURES:

1. Primary Outcome: Physician Follow up
Description: Results reflect the count of participants who were seen by an ophthalmologist for follow-up care within 6 months of their recommended appointment time, and those who did not attend the scheduled follow-up appointment.
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Personalized eHealth Education & Motivational Interviewing | Standard Education
Number analyzed (Participants) | 247 | 243
Participants
  Adherent to recommended follow up | 150 | 144
  Not Adherent to recommended follow up | 97 | 99
Statistical Analysis 1: Comparison: Personalized eHealth Education & Motivational Interviewing vs Standard Education; Test type: Other; p = 0.7399, Chi-squared

ADVERSE EVENTS:
Description: Adverse event data was not collected within the context of the educational trial because the intervention (personalized education and coaching) vs. control (standard education) were so low risk.
Arm/Group | Personalized eHealth Education & Motivational Interviewing | Standard Education
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT04274764/Prot_000.pdf
  • Informed Consent Form (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT04274764/ICF_001.pdf